CLINICAL TRIAL: NCT03662737
Title: A Visuomotor Rotation Task as a Biomarker of Cerebellar Dysfunction in Chronic Cannabis Use
Brief Title: VRT as a Biomarker of Cerebellar Dysfunction in Chronic Cannabis Use
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Hugo López-Pelayo, MD, PhD, Head of Addiction Unit, Hospital Clinic of Barcelona
Other Study IDs: TRV-CAN
Record Dates: First submitted 2018-09-03; First posted 2018-09-07 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cannabis Use; Alcohol Use Disorder; Healthy
Keywords: Visuomotor task
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 -Chronic cannabis use: Individuals between 18 and 50 years old who have been using at least 2 joints per day for at least 3 years. They should have used cannabis during the last 24h but not during the 3h prior to participation to the study and they should test positive for cannabis in their urine. Individuals with another substance use or severe mental disorder will be excluded (except tobacco use)
  Interventions: Diagnostic Test: Visuomotor adaptation task
- Group 2 - Alcohol dependence: Individuals between 18 and 50 years old diagnosed with alcohol use disorder according to DSM-V criteria and have been consuming alcohol for at least 3 years. Individuals who are diagnosed with another substance use or severe mental disorder will be excluded (except tobacco use).
  Interventions: Diagnostic Test: Visuomotor adaptation task
- Control Group: Individuals matched in gender and age with the experimental groups and with no diagnosis of substance use or severe mental disorder (except tobacco use)
  Interventions: Diagnostic Test: Visuomotor adaptation task

INTERVENTIONS:
Diagnostic Test: Visuomotor adaptation task — We will measure performance of the subjects of each group on the visuomotor adaptation task, especially in the rotation condition, in which a perturbation will be induced between the anticipated location of the hand and the provided visual feedback, and in the washout condition, in which the rotation will be removed. We expect that subjects with cannabis use disorder will not show the expected implicit motor adaptation to the perturbation and consequently no deterioration of performance on the task, due to cannabis-induced cerebellar damage. In other words, we want to show that this visuomotor task is a cheap and quick biomarker of cerebellar dysfunction in chronic cannabis users.

SUMMARY:
Chronic cannabis consumption has been associated with poor psychosocial functioning that could be associated to cerebellar dysfunction. The cerebellum has a relevant role in adaptation processes and has a high density of cannabinoid 1 receptor (CB1R). Implicit motor learning is a cerebellum dependent function that can be measured with a visuomotor rotation task (VRT).

The project aims to identify a sensitive and specific biomarker of cerebellum dysfunction in chronic cannabis users. The investigators would like to demonstrate that the visuomotor rotation paradigm is valid to measure and quantify such a dysfunction.

A longitudinal prospective study with a 3 month follow-up is proposed. 3 groups will be included: 1) chronic cannabis users; 2) individuals with an alcohol use disorder; and 3) healthy controls. All groups will be matched by sex and age. Forty individuals will be included in each group. Individuals will be assessed at baseline, at first month and at 3-months of follow-up. Sociodemographic and clinical data will be recorded. Information on cannabis consumption will be registered using an App.

Participants will do the visuomotor rotation task and answer three questionnaires: the Intrinsic Motivation Inventory, the Scale for the assessment and rating of ataxia (SARA) and the Harris tests for lateral dominance.

The biomarker developed by this project will facilitate the detection of cerebellar alterations in chronic cannabis users, and will permit to quantify and monitor such alteration over time. The team's intention is to patent the proposed model and disseminate it in order to use it in clinical practice at both primary and specialized health centres.

DETAILED DESCRIPTION:
The subjects have to realize movements towards a target, at a digitizing tablet, holding a digitizing pencil. Visual feedback is projected on a screen surface in front of the subject, which hides the sight of actual movements from the latter. In the experimental condition of rotation, the experimenter introduces a rotation of 45 grades between the movement realized by the subject and the visual feedback that is provided on the screen. Then, the subject is provided with a strategy in order to overcome this perturbation: that is, to make the movement aiming 45 grades to the opposite direction from the introduced rotation. This explicit strategy leads to immediate correction of the error, but as the time passes subjects tend to commit more and more errors due to implicit motor adaptation. This happens because the motor control system tends to correct the perceived perturbation between the anticipated and the actual location of the hand in an automatic and unconscious way. The conflict between the implicit and explicit strategies has the surprising consequence of a persistent and accumulative deterioration of performance that can only be resolved when the participants abandon the explicit strategy. Subjects with cerebellar damage show deficits in implicit motor learning and for this reason they do not show this progressive deterioration of performance. Given that chronic cannabis abuse can lead to cerebellar damage, the investigators hypothesize that subjects from the experimental group 1 (cannabis use) will have a significant smaller directional error on the rotation condition than controls. A second hypothesis is that this effect will be cannabis-specific, due to the high CB1R concentration on the cerebellum, so the alcohol dependence group is expected to perform similarly to control group

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* Right-handed
* Daily consumption of cannabis for at least 2 years (cannabis group) or diagnosed Alcohol Use Disorder (alcohol group)

Exclusion Criteria:

* Non-corrected visual deficits
* Regular consumption of other drugs except nicotine
* Other Axis I or neurological diagnosis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The experimental group 1 (cannabis use) will consist of the patients of the Addiction Unit of Hospital Clinic that are seeking or already are in treatment for cannabis use or participants that fulfil the eligibility criteria and contact the responsible for this study investigators , after the diffusion of the study. The experimental group 2 (alcohol use) will consist of patients of the Addiction Unit of Hospital Clinic that are in treatment for alcohol dependency. The control subjects will be recruited through the public diffusion of the study.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in directional error between baseline and after cessation of cannabis use | The visuomotor adaptation task duration will not exceed 20 minutes and subjects are expected to realize it at three different time points: baseline, 1 month, 3 months
  Directional error of hand movement trajectories towards the target object on the rotation condition of the visuomotor rotation task.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Gual, MD,PhD, Principal Investigator — Hospital clinic Bracelona
Locations (1):
- Hospital Clínic, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hall W, Degenhardt L. Adverse health effects of non-medical cannabis use. Lancet. 2009 Oct 17;374(9698):1383-91. doi: 10.1016/S0140-6736(09)61037-0. PMID 19837255
- [Background] Moore TH, Zammit S, Lingford-Hughes A, Barnes TR, Jones PB, Burke M, Lewis G. Cannabis use and risk of psychotic or affective mental health outcomes: a systematic review. Lancet. 2007 Jul 28;370(9584):319-28. doi: 10.1016/S0140-6736(07)61162-3. PMID 17662880
- [Background] Silins E, Horwood LJ, Patton GC, Fergusson DM, Olsson CA, Hutchinson DM, Spry E, Toumbourou JW, Degenhardt L, Swift W, Coffey C, Tait RJ, Letcher P, Copeland J, Mattick RP; Cannabis Cohorts Research Consortium. Young adult sequelae of adolescent cannabis use: an integrative analysis. Lancet Psychiatry. 2014 Sep;1(4):286-93. doi: 10.1016/S2215-0366(14)70307-4. Epub 2014 Sep 10. PMID 26360862
- [Background] Batalla A, Bhattacharyya S, Yucel M, Fusar-Poli P, Crippa JA, Nogue S, Torrens M, Pujol J, Farre M, Martin-Santos R. Structural and functional imaging studies in chronic cannabis users: a systematic review of adolescent and adult findings. PLoS One. 2013;8(2):e55821. doi: 10.1371/journal.pone.0055821. Epub 2013 Feb 4. PMID 23390554
- [Background] Lorenzetti V, Solowij N, Yucel M. The Role of Cannabinoids in Neuroanatomic Alterations in Cannabis Users. Biol Psychiatry. 2016 Apr 1;79(7):e17-31. doi: 10.1016/j.biopsych.2015.11.013. Epub 2015 Dec 4. PMID 26858212
- [Background] Lorenzetti V, Solowij N, Fornito A, Lubman DI, Yucel M. The association between regular cannabis exposure and alterations of human brain morphology: an updated review of the literature. Curr Pharm Des. 2014;20(13):2138-67. doi: 10.2174/13816128113199990435. PMID 23829361
- [Background] Crean RD, Crane NA, Mason BJ. An evidence based review of acute and long-term effects of cannabis use on executive cognitive functions. J Addict Med. 2011 Mar;5(1):1-8. doi: 10.1097/ADM.0b013e31820c23fa. PMID 21321675
- [Background] Bossong MG, Jager G, Bhattacharyya S, Allen P. Acute and non-acute effects of cannabis on human memory function: a critical review of neuroimaging studies. Curr Pharm Des. 2014;20(13):2114-25. doi: 10.2174/13816128113199990436. PMID 23829369
- [Background] Broyd SJ, van Hell HH, Beale C, Yucel M, Solowij N. Acute and Chronic Effects of Cannabinoids on Human Cognition-A Systematic Review. Biol Psychiatry. 2016 Apr 1;79(7):557-67. doi: 10.1016/j.biopsych.2015.12.002. Epub 2015 Dec 8. PMID 26858214
- [Background] Burns HD, Van Laere K, Sanabria-Bohorquez S, Hamill TG, Bormans G, Eng WS, Gibson R, Ryan C, Connolly B, Patel S, Krause S, Vanko A, Van Hecken A, Dupont P, De Lepeleire I, Rothenberg P, Stoch SA, Cote J, Hagmann WK, Jewell JP, Lin LS, Liu P, Goulet MT, Gottesdiener K, Wagner JA, de Hoon J, Mortelmans L, Fong TM, Hargreaves RJ. [18F]MK-9470, a positron emission tomography (PET) tracer for in vivo human PET brain imaging of the cannabinoid-1 receptor. Proc Natl Acad Sci U S A. 2007 Jun 5;104(23):9800-5. doi: 10.1073/pnas.0703472104. Epub 2007 May 29. PMID 17535893
- [Background] Kishimoto Y, Kano M. Endogenous cannabinoid signaling through the CB1 receptor is essential for cerebellum-dependent discrete motor learning. J Neurosci. 2006 Aug 23;26(34):8829-37. doi: 10.1523/JNEUROSCI.1236-06.2006. PMID 16928872
- [Background] Mazzoni P, Krakauer JW. An implicit plan overrides an explicit strategy during visuomotor adaptation. J Neurosci. 2006 Apr 5;26(14):3642-5. doi: 10.1523/JNEUROSCI.5317-05.2006. PMID 16597717
- [Background] Taylor JA, Klemfuss NM, Ivry RB. An explicit strategy prevails when the cerebellum fails to compute movement errors. Cerebellum. 2010 Dec;9(4):580-6. doi: 10.1007/s12311-010-0201-x. PMID 20697860
- [Background] Thames AD, Arbid N, Sayegh P. Cannabis use and neurocognitive functioning in a non-clinical sample of users. Addict Behav. 2014 May;39(5):994-9. doi: 10.1016/j.addbeh.2014.01.019. Epub 2014 Feb 6. PMID 24556155
- [Background] Taylor JA, Krakauer JW, Ivry RB. Explicit and implicit contributions to learning in a sensorimotor adaptation task. J Neurosci. 2014 Feb 19;34(8):3023-32. doi: 10.1523/JNEUROSCI.3619-13.2014. PMID 24553942
- [Background] Stella N. Chronic THC intake modifies fundamental cerebellar functions. J Clin Invest. 2013 Aug;123(8):3208-10. doi: 10.1172/JCI70226. PMID 23863631
- [Background] Prashad S, Filbey FM. Cognitive motor deficits in cannabis users. Curr Opin Behav Sci. 2017 Feb;13:1-7. doi: 10.1016/j.cobeha.2016.07.001. PMID 27482533
- [Background] Bastian AJ. Moving, sensing and learning with cerebellar damage. Curr Opin Neurobiol. 2011 Aug;21(4):596-601. doi: 10.1016/j.conb.2011.06.007. Epub 2011 Jul 5. PMID 21733673